CLINICAL TRIAL: NCT01675037
Title: Hypothalamic-pituitary Effects After Endoscopic Third Ventriculostomy
Status: Terminated | Type: Observational
Why Stopped: Recruitment failure
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 1122602; 2011-A01077-34 (Other: Afssaps)
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Hydrocephalus
Keywords: hypothalamic; pituitary,; endoscopic third ventriculostomy; hydrocephalus
MeSH Terms: conditions — Hydrocephalus; Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood, and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- obstructive: obstructive hydrocephalus in children and adults with biological evaluation
  Interventions: Other: Biological evaluation

INTERVENTIONS:
Other: Biological evaluation — Complete hypothalamic-pituitary hormonal evaluation

SUMMARY:
Background: Endoscopic third ventriculostomy (ETV) is a standard procedure for the treatment of obstructive hydrocephalus in children and adults. Perforation of the third ventricle floor which is part of the hypothalamic-pituitary neuronal network is the key of this surgical procedure.

Purpose: There are no prospective data available about the endocrine effects after ETV in children and adults. The principal aim of this prospective study is to evaluate the variability of hypothalamic-pituitary hormones and clinical effects in children and adults after ETV in order to plan a multicentric study.

DETAILED DESCRIPTION:
Introduction Endoscopic third ventriculostomy (ETV) is a standard procedure for the treatment of obstructive hydrocephalus in children and adults. Perforation of the third ventricle floor which is part of the hypothalamic-pituitary neuronal network is the key of this surgical procedure. Single patients with endocrine or electrolyte abnormalities after ETV have been reported in children or adults. So far there are no prospective data available about the endocrine effects after ETV.

Materials and methods 40 patients (10 children, 30 adults) with obstructive hydrocephalus and inclusion criteria will undergo ETV in our neurosurgical department. Complete hypothalamic-pituitary hormonal evaluation will be done, in children and adults, before the procedure and at 3 and 12 month after ETV. At 3 month, a brain MRI, with hypothalamic-pituitary specifics sequences, will be performed and compared to the preoperative one. Follow up will be at 3 and 12 month after ETV.

Interventions: ETV is performed under general anesthesia with a rigid endoscope. Perforation is made just behind the clivus, halfway between the infundibulum and the mammillary bodies in the midline using a monopolar electrode, followed by dilatation with an inflated balloon catheter. In our department, this procedure is performed only by 2 senior surgeons.

Number of subjects: 40 patients: 10 children, 30 adults. Statistical analysis: stratified analysis.

ELIGIBILITY:
Inclusion Criteria:

* all patients over 6 months old with obstructive hydrocephalus who are referred for planned endoscopic third ventriculocisternostomy

Exclusion Criteria:

* MRI contraindication, non obstructive hydrocephalus, life expectancy inferior of 3 months, ETV in emergency, hydrocephalus aetiology interaction with hypothalamic-pituitary hormones, hydrocephalus already treated, basilar artery malformations, to be allergic to tetracosactide (synacthene) and to benserazide (Levodopa).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients over 6 months-old with obstructive hydrocephalus who are referred for planned endoscopic third ventriculocisternostomy to department of neurosurgery in University Hospital of Toulouse, France.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Variability of hypothalamic-pituitary hormones after endoscopic third ventriculostomy | 12 months
  Complete hypothalamic-pituitary hormonal evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Franck-Emmanuel Roux, MD,PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Univesity Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No